CLINICAL TRIAL: NCT05949684
Title: A Phase 3, Open-label, Randomized Study to Compare the Efficacy and Safety of Luspatercept (ACE-536) vs Epoetin Alfa for the Treatment of Anemia Due to Revised International Prognostic Scoring System (IPSS-R) Very Low, Low, or Intermediate-Risk Myelodysplastic Syndrome (MDS) in Erythropoiesis-Stimulating Agent (ESA)-Naive Participants Who Are Non-Transfusion Dependent (NTD): The "ELEMENT-MDS" Trial
Brief Title: ELEMENT-MDS: A Study to Compare the Efficacy and Safety of Luspatercept in Participants With Myelodysplastic Syndrome (MDS) and Anemia Not Receiving Blood Transfusions
Acronym: ELEMENT-MDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA056-025; 2022-500430-29-00 (Other: EU CTR Number)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Luspatercept; BMS-986346; ACE-536; Myelodysplastic Syndrome; Epoetin alfa; Erythropoietin stimulating agent (ESA); Myelodysplastic Syndromes (MDS); Anaemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Luspatercept (Experimental)
  Interventions: Biological: Luspatercept
- Epoetin Alfa (Active Comparator)
  Interventions: Biological: Epoetin Alfa

INTERVENTIONS:
Biological: Luspatercept — Specified dose on specified days
  Other Names: BMS-986346; ACE-536; Reblozyl®
  Arms: Luspatercept
Biological: Epoetin Alfa — Specified dose on specified days
  Other Names: Epogen®; PROCRIT®; BINOCRIT
  Arms: Epoetin Alfa

SUMMARY:
The purpose of the study is to compare the efficacy and safety of Luspatercept vs epoetin alfa in the treatment of anemia in adults due to IPSS-R very low, low, intermediate-risk MDS in ESA-naïve participants who are non-transfusion dependent (NTD).

ELIGIBILITY:
Inclusion Criteria

* Participant has documented diagnosis of MDS according to World Health Organization (WHO) 2016 that meet IPSS-R classification of very low, low, or intermediate-risk disease, (intermediate-risk of ≤ 3.5 IPSS-R score) confirmed via bone marrow aspirate and:.

  i) < 5% blasts in bone marrow and < 1% blasts in peripheral blood.
* Participant is not transfusion dependent (NTD) based on IWG2018 criteria.
* Participant is erythropoiesis-stimulating agent naive. Participants may be randomized at the investigator's discretion if the participant received no more than 2 prior doses of epoetin alfa, epoetin alfa biosimilar, or darbepoetin alfa, with the last dose at least 8 weeks prior to randomization.
* Participant has a baseline endogenous serum erythropoietin (sEPO) level of ≤ 500 U/L.
* Participant has symptoms of anemia:.

  i) Participant records a severity score of "moderate" or greater on at least 1 PGI-S item of fatigue, weakness, shortness of breath, or dizziness performed during the screening period.
* Participant has a baseline Hb concentration prior to randomization of ≤ 9.5 g/dL. The baseline Hb will be calculated using the mean of the two lowest available Hb measurements within 16 weeks prior to randomization and must include at least one central lab Hb reading done within the screening period (no more than 35 days before randomization). The two Hb measurements must have been performed at least seven days apart. Hb levels less than 21 days following RBC transfusion should not be used. Split samples for local assessments are not required.

Exclusion Criteria

* Participant with secondary MDS (that is, MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases).
* Participant with known history of diagnosis of AML.
* Participant with history of cerebrovascular accident (including ischemic, embolic, and hemorrhagic cerebrovascular accident), transient ischemic attack, deep venous thrombosis (including proximal and distal), pulmonary or arterial embolism, arterial thrombosis, or other venous thrombosis within 6 months prior to randomization.
* Participant with a history of pure red cell aplasia and/or antibody against erythropoietin.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2030-03-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with lower-risk non-transfusion dependent myelodysplastic syndromes (NTD-MDS) who converted to Transfusion Dependence (TD) during any continuous 16-week interval within the 96-week treatment period | Up to Week 96
  TD is defined as ≥ 3 red blood cells (RBC) units/16 weeks assessed by International Working Group (IWG) 2018.

SECONDARY OUTCOMES:
Number of participants with an increase from baseline in mean Hb values of ≥ 1.5 grams/deciliter (g/dL) in any continuous 16-week interval within the 48 week Treatment Period in the absence of transfusion | Up to Week 48
Number of participants with an increase from baseline in mean Hb values of ≥ 1.5 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | Up to Week 48
Number of participants with an increase from baseline in mean Hb values of ≥ 1.5 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | From Week 49 to Week 96
Number of participants with an increase from baseline in mean Hb values of ≥ 1.5 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | Up to Week 96
Number of participants with an increase from baseline in mean Hb values of ≥ 1.0 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | Up to Week 48
Number of participants with an increase from baseline in mean Hb values of ≥ 1.0 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | From Week 49 to Week 96
Number of participants with an increase from baseline in mean Hb values of ≥ 1.0 g/dL in any continuous 24-week interval within the 48-week and 96-week treatment period in the absence of transfusion | Up to Week 96
Mean Hb change over fixed 24-week periods compared to the baseline Hb | Baseline, Week 24, Week 48, Week 72, Week 96
Number of participants with an increase from baseline in mean Hb values of ≥ 1.5 g/dL in any continuous 16-week interval within the 96-week treatment period in the absence of transfusion | Up to Week 96
Number of participants with TD by week 48 | Up to Week 48
Time to TD (IWG 2018 defined as ≥ 3 RBC units/16 weeks) during any continuous 16-week interval until the end of study | Up to 5 years
Time from first Luspatercept dose to first RBC transfusion | Up to 5 years
Duration of median hematologic improvement in erythroid response(mHI-E) in participants with an increase from baseline in mean Hb values of ≥1.5g/dL in any continuous 16-week interval within 48-week treatment period in absence of transfusion | Up to Week 48
Duration of median hematologic improvement in erythroid response(mHI-E) in participants with an increase from baseline in mean Hb values of ≥1.5g/dL in any continuous 16-week interval within 96-week treatment period in absence of transfusion | Up to Week 96
Time from first dose to first day of response (increase in mean Hb values of ≥ 1.5 g/dL in any continuous 16-week interval within the 48-week Treatment Period in the absence of transfusion) | Up to Week 48
Time from first dose to first day of response (increase in mean Hb values of ≥ 1.5 g/dL in any continuous 16-week interval within the 96-week Treatment Period in the absence of transfusion) | Up to Week 96
Number of participants with RBC transfusion independence over at least a consecutive 24-week period | Up to 5 years
Number of transfusions | Up to 5 years
Number of transfusions visits/units | Up to 5 years
Change from baseline in subscales of self-reported health-related quality-of-life (HRQoL) assessed by the Functional Assessment of Cancer Therapy - Anemia (FACT-An) | Baseline, Up to 5 years
Change from baseline in self-reported HRQoL assessed by the European quality of life questionnaire 5-dimension (EQ-5D-5L) | Baseline, Up to 5 years
Number of participants with adverse events (AEs) | Up to Week 102
Number of participants with antidrug antibody (ADA) (positive or negative) | Up to Week 102
Pharmacokinetics (PK): Serum concentration | Up to Week 96
PK: Area under the plasma concentration time curve (AUC) | Up to Week 96
Number of participants with a platelet response at Week 24, Week 48 and Week 96 | Up to Week 96
  Platelet response is defined as an increase from baseline in number of platelets to ≥ 30 × 10^9/L at Week 24, Week 48 and Week 96.
Number of participants with a neutrophil response at Week 24, Week 48 and Week 96 | Up to Week 96
  Neutrophil response is defined as an absolute increase from baseline of > 0.5 × 10^9/L neutrophils at Week 24, Week 48 and Week 96.
Number of participants with acute myeloid leukemia (AML) progression | Up to 5 years
Time to AML progression | Up to 5 years
Number of participants with high risk myelodysplastic syndromes (MDS) progression | Up to 5 years
Time to high-risk MDS progression | Up to 5 years
Time from date of randomization up to death due to any cause | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (169):
- United States (39):
  - Community Cancer Institute, Clovis, California
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - Local Institution - 0095, Fresno, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 120), Los Angeles, California
  - St. Joseph Hospital, Orange, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - John Muir Health - Behring Pavilion, Walnut Creek, California
  - Local Institution - 0098, Fort Collins, Colorado
  - Hartford Hospital (HH), Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Halifax Health Medical Center, Daytona Beach, Florida
  - Local Institution - 0230, Daytona Beach, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Local Institution - 0224, Margate, Florida
  - BRCR Global, Plantation, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Advanced Research, Tamarac, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0240, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Northwest Cancer Centers, P.C., Dyer, Indiana
  - Local Institution - 0232, Pikeville, Kentucky
  - Our Lady of the Lake RMC, Baton Rouge, Louisiana
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Local Institution - 0097, New Orleans, Louisiana
  - American Oncology Partners, PA, Bethesda, Maryland
  - Metro-Minnesota Community Clinical Oncology, Saint Louis Park, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - VCU Health Adult Outpatient Pavillion, Richmond, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Local Institution - 0213, Seattle, Washington
- Argentina (3):
  - Centro Medico Barrio Parque, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Británico de Buenos Aires, Buenos Aires
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Pindara Private Hospital, Gold Coast, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
- Brazil (4):
  - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - HEMORIO, Rio de Janeiro
  - Hospital das Clinicas FMUSP, São Paulo
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Chile (4):
  - Enroll SpA, Santiago, Santiago Metropolitan
  - FALP, Santiago, Santiago Metropolitan
  - Clínica Inmunocel, Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (25):
  - Local Institution - 0109, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Local Institution - 0223, Chongqing, Chongqing Municipality
  - Local Institution - 0096, Fuzhou Fujian, Fujian
  - Local Institution - 0220, Xiamen, Fujian
  - Local Institution - 0031, Guangzhou, Guangdong
  - The Second Afilliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Harbin, Harbin, Heilongjiang
  - People's Hospital of Henan Province, Zhengzhou, Henan
  - Local Institution - 0108, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Local Institution - 0043, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shaanxi provincial people's hospital, Xi’an, Shanxi
  - Local Institution - 0075, Chengdu, Sichuan
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Local Institution - 0281, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Colombia (4):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Sociedad De Oncologia Y Hematologia Del Cesar, Valledupar, Cesar Department
  - Fundación Cardiovascular de Colombia, Piedecuesta, Santander Department
  - Oncomédica S.A.S, Montería
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (9):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours, Indre-et-Loire
  - Chu Grenoble Alpes, La Tronche, Isère
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Hôpital Saint-Louis, Paris
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse
- Germany (12):
  - Local Institution - 0261, Erding, Bavaria
  - Local Institution - 0250, Kempten (Allgäu), Bavaria
  - Gemeinschaftspraxis für Hämatologie und Onkologie Münster, Münster, North Rhine-Westphalia
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
  - Praxis fur Hamatologie und Onkologie, Berlin
  - Local Institution - 0028, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Local Institution - 0255, Lübeck
  - Kliniken Ostalb, Stauferklinikum, Mutlangen
  - Gemeinschaftspraxis Dres. med. Björn Schöttker & Dominik Pretscher, Würzburg
- Greece (6):
  - Local Institution - 0242, Pátrai, Achaḯa
  - University Hospital of Patras, Pátrai, Achaḯa
  - University General Hospital of Alexandroupoli, Alexandroupoli, Anatolikí Makedonía Kai Thráki
  - General Hospital of Athens "G. Gennimatas", Athens, Attikí
  - General Hospital of Athens "Laiko", Athens, Attikí
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
- Local Institution - 0034, Hksar, Hong Kong
- Hungary (3):
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet, Eger, Heves County
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem, Budapest
- India (8):
  - Hemato Oncology Clinic, Ahmedabad, Gujarat
  - Local Institution - 0273, Ahmedabad, Gujarat
  - Local Institution - 0177, Bengaluru, Karnataka
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Institute of Medical Sciences and Sum Hospital, Bhubaneswar, Odisha
  - Local Institution - 0185, Hyderabad
  - Local Institution - 0186, New Delhi
- Italy (10):
  - Fondazione Policlinico Tor Vergata, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Grande Ospedale Metropolitano - Presidio Morelli, Reggio Calabria
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Japan (10):
  - Local Institution - 0123, Kitakyushu-shi, Fukuoka
  - Local Institution - 0117, Sapporo, Hokkaido
  - Local Institution - 0126, Amagasaki, Hyōgo
  - Local Institution - 0120, Sagamihara, Kanagawa
  - Local Institution - 0118, Sendai, Miyagi
  - Local Institution - 0125, Ōsaka-sayama, Osaka
  - Local Institution - 0121, Shimotsuga, Tochigi
  - Local Institution - 0124, Nagasaki
  - Local Institution - 0122, Osaka
  - Local Institution - 0119, Tokyo
- Mexico (4):
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Hematológica Alta Especialidad SC, consultorio 830, Huixquilucan
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Unidad Médica Onco-hematológica, Puebla City
- Poland (4):
  - Specjalistyczny Szpital im. dra Alfreda Sokołowskiego w Wałbrzychu, Wałbrzych, Lower Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - MTZ Clinical Research powered by Pratia, Warsaw
- Puerto Rico (2):
  - Auxilio Mutuo Cancer Center, San Juan
  - Local Institution - 0237, San Juan
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital La Princesa, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05949684.html